CLINICAL TRIAL: NCT01634399
Title: An Open-Label, Randomised, 2-Period, 2-Treatment, 2-sequence, Crossover Single-dose Bioequivalence Study of Quetiapine 25 mg Tablet [Test Formulation; Torrent Pharmaceuticals Ltd., India] Versus Seroquel® 25 mg Tablet [Reference Formulation; AstraZeneca, USA] in Healthy Human Volunteers Under Fed Condition.
Brief Title: Bioequivalence Study of Torrent Pharmaceuticals Ltd's Bioequivalence Study of Torrent Pharmaceuticals Ltd's Quetiapine Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PK-08-190
Record Dates: First submitted 2012-06-27; First posted 2012-07-06 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Torrent's Quetiapine Fumarate Tablets

SUMMARY:
Objective:

Primary objective of the present study was to compare the single dose bioequivalence of Torrent's Quetiapine Fumarate Tablets 1 × 25 mg. Dosing periods of the study were separated by a washout period of 7 days.

Study Design:

Open label, Randomized, Two-Way, Crossover, Single-Dose Bioequivalence Study

ELIGIBILITY:
Inclusion Criteria:

The volunteers were included in the study based on the following criteria:

* Sex: male.
* Age: 18 - 45 years.
* Volunteer with BMI of 18-27 (inclusive both) kg/m2 with minimum of 50 kg weight.
* Healthy and willing to participate in the study.
* Volunteer willing to adhere to the protocol requirements and to provide written informed consent.
* Non-smokers or smoker who smokes less than 10 cigarettes per day

Exclusion Criteria:

The volunteers were excluded from the study based on the following criteria:

* Clinically relevant abnormalities in the results of the laboratory screening evaluation.
* Clinically significant abnormal ECG or Chest X-ray.
* Systolic blood pressure less than 100 mm Hg or more than 140 mm Hg and diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
* Pulse rate less than 50/minute or more than 100/minute.
* Oral temperature less than 95°P or more than 98.6°P.
* Respiratory rate less than 12/minute or more than 20/minute
* History of allergy to the test drug or any drug chemically similar to the drug under investigation.
* History of alcohol or drug abuse
* Positive breath alcohol test
* Recent history of kidney or liver dysfunction.
* History of consumption of prescribed medication since last 14 days or OTC medication since last 07 days before beginning of the study.
* Volunteers suffering from any chronic illness such as arthritis, asthma etc.
* History of heart failure.
* HIV, HCV, HBsAg positive volunteers.
* Opiate, tetra hydrocannabinol, amphetamine, barbiturates, benzodiazepines, - - - Cocaine positive volunteers based on urine test.
* Volunteers suffering from any psychiatric (acute or chronic) illness requiring medications.
* Administration of any study drug in the period 0 to 3 months before entry to the study.
* History of significant blood loss due to any reason, including blood donation in the past 3 months.
* History of pre-existing bleeding disorder.
* Existence of any surgical or medical condition, which, in the judgment of the chief investigator and/or clinical investigator/physician, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of volunteers.
* Inability to communicate or co-operate due to language problem, poor mental development or impaired cerebral function.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Bio Evaluation Centre, Torrent Pharmaceuticals Ltd.,, Village Bhat, Gandhinagar, Gujarat, India